CLINICAL TRIAL: NCT02701426
Title: Obesity and Pregnancy : Study of Factors Influencing Participation in a Program Combining Physical Activity and Nutritional Counseling
Brief Title: Obesity & Pregnancy: Factors Influencing Participation in a Physical Activity and Nutritional Counseling Program
Acronym: OGAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of funding granted
Sponsor: University Hospital, Lille (Other)
Collaborators: University of Lille Nord de France (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014_72; 2015-A01085-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Overweight; Pregnancy
Keywords: Macrosomia; Weight gain; Participation; Adhesion; Physical activity; Nutrition
MeSH Terms: conditions — Obesity; Overweight; Weight Gain; Tissue Adhesions; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- participant (Experimental): agree to participate to the program combining physical activity and nutritional counseling
  Interventions: Behavioral: physical activity and nutritional counseling
- no participant (No Intervention): disagree to participate to the program

INTERVENTIONS:
Behavioral: physical activity and nutritional counseling — The program will last 12 weeks, and will include three workshops on diet of the pregnant and lactating women, and the young child. Physical activity sessions will be offered once a week.
  Arms: participant

SUMMARY:
Background:

Obesity increasingly affects young women and contributes to increased maternal, fetal and neonatal complications. Maternal obesity contributes to the subsequent development of childhood obesity not only through social and environmental mechanisms but also through biological processes referring to the original concept of the developmental health and disease. Data suggest that management during pregnancy through nutrition counseling and adequate physical activity will help to break the familial vicious circle of obesity. To help program to be effective it is important to understand the factors that modulate participation. However, few studies have been conducted to assess the determinants that influence participation.

Goal:

The main objective is to analyze 15 factors that influence participation in a program combining physical activity and nutritional counseling among pregnant women with BMI ≥ 25 kg/m2. Secondary objectives are :

* to identify the data that influence adherence and to show that assiduous women will have a better control of weight gain and a reduction of maternal and fetal complications.
* to understand the biological mechanisms involved

Strategy and method:

A prospective research evaluating the participation in an educational program, including nutritional support and adequate physical activity, will be offered to overweight and obese pregnant women. The program will last 12 weeks, and will include three workshops on diet of the pregnant and lactating women, and the young child. Physical activity sessions will be offered once a week. Fifteen independent variables likely to influence participation will be analyzed. The association between participation and the risk of maternal and fetal pregnancy complications related to obesity will be analysed. Meanwhile, more fundamental research will be considered to determine of the biological factors involved.

DETAILED DESCRIPTION:
This is a prospective study that will be conducted in pregnant women with a BMI ≥ 25 kg/m2, aged from 18 to 42 years. Participation in the program will be offered between 12 and 22 + 6 weeks of pregnancy. Women with a history of more than 2 miscarriages, severe heart disease (arrhythmia, previous myocardial infarction), bleeding in the first trimester, multiple pregnancy, unstable thyroid disease, hypertension, diabetes, or any other medical conditions that can interfere with the practice of physical activity during pregnancy will not be allowed to participate in the program for medical reasons. The participants will sign an informed consent. The intervention will be an educational program called "Eat well, move well for to the baby's health," including nutritional counselling and physical activity exercises. The control group will receive usual care as a simple information. The intervention will take place between 24 and 36 weeks of pregnancy. Women will be evaluated before (20-24 weeks gestation (SA)), during the intervention (32-34 SA), and finally 8 weeks after childbirth during the postnatal visit. All patients with benefit from obstetric monitoring according with the French recommendations with a monthly consultation and ultrasonography exams at 22 and 32 wks.

Nutritional support will include 3 workshops of 2 hours within the 12 weeks (one workshop per month). Each workshop session will be conducted in groups of 10 to 15 participants. These workshops will aim firstly to inform patients of weight gain recommendations during pregnancy and food recommendations.

Workshop No. 1 will provide information on the goals of weight gain during pregnancy, and will target the implementation of recommendations in terms of diet during pregnancy. The messages will be specifically adapted to the population of obese women including dietary advices, work on erroneous beliefs and representations, work on the motivation to change eating habits and reduction of the harmful link between emotions and eating. Thus, beyond the information, this workshop will have the primary role to develop a diet suitable for pregnancy in obese women. This workshop will be led by a dietician and psychologist. It will take place between the 1st and 4th week of the program.

Workshop No. 2 will inform the benefits of breastfeeding for the child and the mother (including its impact on weight loss during the postpartum period, especially important in obese women). As in the previous workshop, the objective will be to obtain the application of the recommendations on diet during breastfeeding. The general message will be adapted to the problems specific to obese women: work on the social, educational, family, removal of beliefs and motivational brakes. This workshop will be led by a dietician and a midwife and will take place between the 5th and 8th week of the program.

Workshop No. 3 will target the diet in the postpartum period and nutritional needs of the newborn and young child. Beyond dietary information, specific work will be done on motivation to take care of the body after pregnancy and breastfeeding, and especially the fight against the beliefs of the food needs of the newborn, typically found in obese mothers (fear of missing, hunger equated with suffering, the emotional power as substitute) This workshop will take place between the 9th and 12th week of the program and will be led by a dietician and a pediatric nurse.

The exercise program will feature sessions developed by the North Committee of the French Federation of Physical Education and Voluntary Gymnastics. On the program, which lasts 12 weeks per patient, there will be inputs and outputs permanent in the group based on inclusions. The program will be continued for the duration of the research. This program will propose 3 weekly slots of physical activities so that participants can take at least a weekly session. Ideally they will be encouraged to practice a second session and to perform exercises by their own. The personal session can be a walk on the weekend, or an indoor gym classes in one a club, an aqua fit session ... or exercises proposed by the coach to replicate at home. The participants will be able to record and monitor their practice using the logbook.

Evaluation of the program "Eat well, move well for the baby's health" The investigators will do the assessment before during and after the program. Patients will have a logbook in which they will notice physical activity performed. This book will include questionnaires to complete.

1. Food Evaluation The investigators will use a food behavior questionnaire (18 items) and 5 direct questions for a semi-quantitative assessment (sweet beverages consumption, fat, portion sizes). All these elements for assessing eating behavior (uncontrolled eating, hunger, cognitive restriction), the type of food consumed (carbohydrates, fats and proteins). The evaluation will be conducted by dieticians.
2. Evaluation of physical activity Physical activity of patients will be estimated using the French Physical Activity Questionnaire in Pregnancy (QFAPG). This self administered questionnaire will have a qualitative vision (business type) and quantitative activity through 33 questions on "sports" on "household activities " on "activities at work " and also on "activities related to transportation".

   Physical activity will be quantitatively measured for each patient who will receive an accelerometer (The Actigraph, Manufacturing Technology Inc., model wActisleep +, Pensacola, Florida USA) that will record the intensity of the efforts made during a period of 7 days.
3. Well-being Evaluation Well-being will be evaluated using the positive and negative affect schedule Questionnaire. which is sensitive to changes over time and assesses the positive and negative affects. It will assess the program's impact on the positive / negative affect.

ELIGIBILITY:
Inclusion criteria :

* Overweight and obese pregnant women
* Age from 18 to 45 years old
* Singleton pregnancy between 12+0 to 22+6 weeks of pregnancy

Exclusion criteria:

* History of more than 2 miscarriages
* Severe heart disease (arrhythmias, history of myocardial infarction)
* Multiple pregnancy
* Unstable thyroid disease
* Uncontrolled hypertension
* Pre-gestational diabetes
* Bariatric surgery
* Any medical condition that may interfere with physical activity during pregnancy
* Minor or absence of health insurance
* Trusteeship or tutorship
* Refusal to participate in research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Number of participant that will participate to the program | at 36 weeks of gestation (WG)

SECONDARY OUTCOMES:
Macrosomia / Birth weight | at birth
Gestational weight gain | at birth
Pregnancy complications | between 28 weeks of gestation and term
  Gestational diabetes, gravidic hypertension and preeclampsia
Number of patients with C-section or an instrumental extraction | at birth
  C-section vaginal delivery, instrumental extraction
eating behavior before, during and after the program | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation, within 6-8 weeks post-partum
  Three eating factors questionnaire / semi-qualitative questionnaire
Questionnaire of physical activity | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation, within 6-8 weeks post-partum
  french questionnaire of physical activity
Questionnaire for self-esteem | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation, within 6-8 weeks post-partum
  Positive and Negative Affect Schedule (PANAS) questionnaire
number of neonates with neonatal trauma | at birth
  fractures, shoulder dystocia, brachial plexus injury
Apgar score | at birth
Arterial umbilical pH | at birth
number of neonates with hyperbilirubinemia | Within 7 days after birth
  total serum bilirubin level > 86 micro mol/L
Number of neonates needing intensive care transfer | Within 7 days after birth
Neonatal adiposity | at birth
  measurement of shoulder fat thickness in mm
Maternal weight | within 6-8 weeks post-partum
Infant weight | within 6-8 weeks post-partum
duration of Breastfeeding | within 6-8 weeks post-partum
  in weeks
Maternal Plasmatic cholesterol levels before, during and after the program | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
Maternal Plasmatic leptin levels | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
maternal plasmatic glycemic levels | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
microRNA levels in maternal milk | 2 or 3 days after birth
Physical activity measured with accelerometers | between 32 and 34 Weeks of gestation and within 6-8 weeks post-partum
  measurements for 1 week
Maternal Plasmatic triglyceride levels before, during and after the program | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
Maternal Plasmatic Apolipoprotein levels before, during and after the program | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
Maternal plasmatic apelin levels | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
maternal plasmatic insulin levels | between 20-24 weeks of gestation, between 32 and 34 weeks of gestation and at birth
Pittsburgh Sleep Quality Index | during 7 days between 20-24 weeks of gestation, between 32 and 34 weeks of gestation, within 6-8 weeks post-partum
  is a self-report questionnaire that assesses sleep quality over a 1-month time interval.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Deruelle, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Jeanne de Flandres, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deruelle P. [Obesity and pregnancy]. Gynecol Obstet Fertil. 2011 Feb;39(2):100-5. doi: 10.1016/j.gyobfe.2010.12.001. Epub 2011 Feb 12. French. PMID 21317009
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Derived] Lelorain S, Deruelle P, Behal H, Machet E, Thiblet M, Lengagne-Piedbois C, Deken-Delannoy V, Pigeyre M. Factors influencing participation and regular attendance in a program combining physical activity and nutritional advice for overweight and obese pregnant women. BMC Pregnancy Childbirth. 2024 Jun 28;24(1):449. doi: 10.1186/s12884-024-06648-z. PMID 38943053